CLINICAL TRIAL: NCT02730936
Title: Feasibility Study of the Antimicrobial Hernia Repair Device for Repair of Ventral or Incisional Hernia
Brief Title: Antimicrobial Hernia Repair Device
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision to discontinue the study.
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-12
Record Dates: First submitted 2016-03-30; First posted 2016-04-07 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Ventral Hernias; Incisional Hernias
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Antimicrobial Hernia Repair Device (Experimental): Antimicrobial hernia repair device for repair of ventral or incisional hernias in Class II and III surgical fields.
  Interventions: Device: Antimicrobial Hernia Repair Device

INTERVENTIONS:
Device: Antimicrobial Hernia Repair Device — hernia repair

SUMMARY:
This prospective early feasibility clinical study will collect information regarding the safety and efficacy of the Cook® Antimicrobial Hernia Repair Device to reinforce soft tissue during ventral or incisional hernia repair in clean-contaminated and contaminated (i.e., Class II and Class III) surgical fields.

ELIGIBILITY:
Inclusion Criteria:

* Patient with ventral or incisional hernia that is to be surgically corrected in a Class II and Class III surgical field.

Exclusion Criteria:

* Less than 21 years old
* Unwilling or unable to sign and date the informed consent
* Pregnant, breastfeeding, or planning to become pregnant prior to completing the study
* Unable or unwilling to comply with follow-up schedule
* Simultaneously participating in another investigational drug or device study.
* Medical condition or disorder that would limit life expectancy to less than the primary clinical study endpoint.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01-12 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients that develop a surgical site infection | 6 months
  Surgical site infections (SSI) that will be included in this outcome measure are deep incisional, organ/space, and superficial incisional.

SECONDARY OUTCOMES:
Number of hernia recurrences | 24 months
  Hernia recurrences is the protrusion of abdominal tissue through a defect in the abdominal wall at the site of the hernia repaired during the index procedure.
Frequency of procedural and post-operative adverse events | 24 months
  The adverse events will be bowel erosion, bowl obstruction, delayed wound infection, fever, fistula formation, graft contraction, hernia recurrence, ileus, need for revision/resurgery, pain, premature degradation, wound dehiscence, and other wound complications.